CLINICAL TRIAL: NCT03837899
Title: Phase I/II, Open-Label Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of Durvalumab Monotherapy or in Combination With Tremelimumab in Pediatric Patients With Advanced Solid Tumors and Hematological Malignancies.
Brief Title: Durvalumab and Tremelimumab for Pediatric Malignancies
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D419EC00001; 2018-003118-42 (EudraCT Number)
Record Dates: First submitted 2019-01-24; First posted 2019-02-12 (Actual); Results first posted 2024-03-19 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Pediatric Cancer; Solid Tumor Pediatric; Hematological Malignancies
Keywords: Pediatric, solid tumors, hematological malignancies, durvalumab, tremelimumab, immunotherapy
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Durvalumab / Tremelimumab Combination Therapy (Experimental): Part 1 (dose finding) Durvalumab + tremelimumab Combination Treatment. Durvalumab and tremelimumab are initially administered at dose level 1 and dose escalated based on results from PK modeling and tolerance to determine the RP2D. Both drugs are administered every 4 weeks as intravenous infusions. Tremelimumab is only administered with durvavalumab for 4 doses, from cycles 2-5. (sarcoma, NB and NHL)
  Part 2 (dose expansion phase) Durvalumab + tremelimumab Combination Treatment. Durvalumab and tremelimumab are administered at the RP2D, every 4 weeks as intravenous infusions. Tremelimumab is only administered with durvalumab for 4 doses, from cycles 1-4. Tremelimumab may be added for 4 doses at time of progressive disease. Cohorts: solid tumors, sarcomas, NHL restricted to PMBCL and ALCL subtypes)
  Interventions: Drug: Durvalumab / Tremelimumab Combination Therapy

INTERVENTIONS:
Drug: Durvalumab / Tremelimumab Combination Therapy — Starting dose:
  durvalumab: 20mg/kg tremelimumab: 1mg/kg at cycles 2 to 5 only co-administered with durvalumab. The Recommended Phase 2 dose will be used for the dose expansion phase.
  Other Names: durvalumab: Imfinzi, MEDI4736; tremelimumab: CP-675,206

SUMMARY:
The purpose of the study is to determine the recommended dose of durvalumab and tremelimumab (immunotherapy drugs) in pediatric patients with advanced solid and hematological cancers and expand in a second phase to test the efficacy of these drugs once this dose is determined.

DETAILED DESCRIPTION:
This is a first time in pediatrics study primarily designed to evaluate the safety and tolerability of durvalumab and durvalumab in combination with tremelimumab at increasing doses in pediatric patients with advanced solid malignancies and hematological malignancies (including lymphomas) and for whom no standard of care treatments exist. Although treatment efficacy is not a primary objective of this study given its early phase nature, the patients screened for this study have no curative options and this study offers the potential of some benefit.

The study will also characterize the PK of durvalumab and durvalumab in combination with tremelimumab in children and adolescents and explore potential biological activity and immunogenicity by assessing pharmacodynamics, anti drug antibody (ADA) levels, and anti-tumor activity. The results from this trial will form the basis for decisions for potential future pediatric studies

ELIGIBILITY:
Inclusion Criteria:

* Max Age =17 years
* Solid Tumors (except primary central nervous system malignant tumors): Patients must have a histopathologic confirmation of malignancy. Patients must have progressed or are refractory to standard therapies, and for whom no standard of care treatments exist
* Non-Hodgkin's Lymphoma, limited to primary mediastinal B-cell lymphoma and anaplastic large cell lymphoma. Patients must have progressed or are refractory to standard therapies, and for whom no standard of care treatments exist.
* Provision of diagnostic tumor sample mandated if available
* Evaluable disease
* No prior exposure to immune-mediated therapy
* Adequate organ and marrow function
* Life expectancy of at least 3 months

Exclusion Criteria:

* History of allogeneic organ transplantation (exceptions may be allowed for NHL after discussion with Sponsor). History of autologous bone marrow transplant may be allowed (after discussion with Sponsor).
* Active or prior documented autoimmune or inflammatory disorders (exceptions)
* Uncontrolled intercurrent illness
* History of primary immunodeficiency
* Active infection including tuberculosis, hepatitis B, C or HIV
* Any unresolved toxicity NCI CTCAE version 5.0 Grade ≥2 from previous anticancer therapy (exceptions)

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2024-12-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Gupta, MD, PhD, Study Director — AstraZeneca Global Medicines Development, Academy House
Locations (19):
- United States (5):
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, New Hyde Park, New York
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Charleston, South Carolina
- France (3):
  - Research Site, Lille
  - Research Site, Marseille
  - Research Site, Paris
- Research Site, Cologne, Germany
- Italy (4):
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Rome
  - Research Site, Torino
- Research Site, Utrecht, Netherlands
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Madrid
- United Kingdom (3):
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Study Protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419EC00001&attachmentIdentifier=22d183cf-55ee-4e24-949c-5fdea2f8f4a9&fileName=CSP_redacted.pdf&versionIdentifier=
- See also: CSR Synopsis Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419EC00001&attachmentIdentifier=0f771b05-0335-4531-8f9d-bf150dd375c5&fileName=CSR_synopsis_redacted.pdf&versionIdentifier=
- See also: SAP Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419EC00001&attachmentIdentifier=71e869ee-f7bb-41d8-9d08-ba49c7da3316&fileName=SAP_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This open-label study was conducted in 2 sequential phases: a dose-finding phase (Phase I), followed by a dose-expansion phase (Phase II) in pediatric participants with advanced solid tumors, including sarcoma. Here, results for data analyzed through data cut-off date (DCO) 20-Apr-2023 have been reported.
Pre-assignment Details: Each treatment cycle was 28 days. Overall, 33 participants were enrolled in dose-finding phase and 29 participants were administered study treatment. In dose-expansion phase, 23 participants were enrolled and 21 participants were administered study treatment.
Groups:
- Arm A (>= 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg: Participants who weighed >= 35 kilograms (kg) were administered durvalumab 20 milligram (mg)/kg intravenously (IV) in Cycle 1 followed by durvalumab in combination with tremelimumab 1 mg/kg IV in Cycles 2-5 every 28 days. From Cycle 6 onwards participants were administered durvalumab 20 mg/kg every 28 days until clinical or confirmed disease progression or until any of other discontinuation criterion was met, whichever occurred first.
- Arm A (>= 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg: Participants who weighed >= 35 kg were administered durvalumab 30 mg/kg IV in Cycle 1 followed by durvalumab in combination with tremelimumab 1 mg/kg IV in Cycles 2-5 every 28 days. From Cycle 6 onwards participants were administered durvalumab 20 mg/kg every 28 days until clinical or confirmed disease progression or until any of other discontinuation criterion was met, whichever occurred first.
- Arm B (< 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg: Participants who weighed < 35 kg were administered durvalumab 20 mg/kg IV in Cycle 1 followed by durvalumab in combination with tremelimumab 1 mg/kg IV in Cycles 2-5 every 28 days. From Cycle 6 onwards participants were administered durvalumab 20 mg/kg every 28 days until clinical or confirmed disease progression or until any of other discontinuation criterion was met, whichever occurred first.
- Arm B (< 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg: Participants who weighed < 35 kg were administered durvalumab 30 mg/kg IV in Cycle 1 followed by durvalumab in combination with tremelimumab 1 mg/kg IV in Cycles 2-5 every 28 days. From Cycle 6 onwards participants were administered durvalumab 20 mg/kg every 28 days until clinical or confirmed disease progression or until any of other discontinuation criterion was met, whichever occurred first.
- SARCOMA: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg: Participants with osteosarcoma and Ewing sarcoma, rhabdomyosarcoma, non rhabdomyosarcoma soft tissue sarcoma, and other sarcomas were included in this arm. Participants were administered durvalumab 30 mg/kg IV in combination with tremelimumab 1 mg/kg IV in Cycles 1-4 every 28 days. From Cycle 5 onwards participants were administered durvalumab 30 mg/kg every 28 days until clinical or confirmed disease progression or until any of other discontinuation criterion was met, whichever occurred first.
- STO: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg: Participants with solid tumor other (STO) were included in this arm. Participants were administered durvalumab 30 mg/kg IV in combination with tremelimumab 1 mg/kg IV in Cycles 1-4 every 28 days. From Cycle 5 onwards participants were administered durvalumab 30 mg/kg every 28 days until clinical or confirmed disease progression or until any of other discontinuation criterion was met, whichever came occurred first.
Period: Overall Study
Arm/Group | Arm A (>= 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm A (>= 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | SARCOMA: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | STO: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Started | 7 | 11 | 3 | 8 | 11 | 10
Completed | 1 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 11 | 3 | 8 | 11 | 10
Not completed — Death | 6 | 8 | 3 | 7 | 8 | 7
Not completed — Moved to post-trial access program | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Study specific discontinuation criteria | 0 | 1 | 0 | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Population: The Full analysis set (FAS) included all participants who were assigned to treatment and received at least 1 dose of study treatment.
Groups:
- Arm A (>= 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg: Participants who weighed >= 35 kg were administered durvalumab 20 mg/kg IV in Cycle 1 followed by durvalumab in combination with tremelimumab 1 mg/kg IV in Cycles 2-5 every 28 days. From Cycle 6 onwards participants were administered durvalumab 20 mg/kg every 28 days until clinical or confirmed disease progression or until any of other discontinuation criterion was met, whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | Arm A (>= 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm A (>= 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | SARCOMA: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | STO: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | Total
Number analyzed (Participants) | 7 | 11 | 3 | 8 | 11 | 10 | 50
Age, Customized [Count of Participants; unit: Participants]
  In utero | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Preterm newborn infants (gestational age < 37 weeks) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Newborns (0-27 days) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Infants and toddlers (28 days-23 months) | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Children (2-11 years) | 0 | 5 | 3 | 6 | 7 | 3 | 24
  Adolescents (12-17 years) | 6 | 6 | 0 | 2 | 4 | 7 | 25
  Adults (18-64 years) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  From 65-84 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  85 years and above | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 8 | 1 | 3 | 6 | 5 | 26
  Male | 4 | 3 | 2 | 5 | 5 | 5 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1 | 1 | 0 | 1 | 0 | 0 | 3
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 1 | 0 | 0 | 1 | 1 | 3
  White | 5 | 8 | 2 | 4 | 8 | 6 | 33
  Other | 1 | 1 | 1 | 3 | 1 | 3 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 1 | 1 | 0 | 2 | 7
  Not Hispanic or Latino | 6 | 9 | 2 | 7 | 11 | 8 | 43

OUTCOME MEASURES:

1. Primary Outcome: Dose-Finding Phase: Maximum Serum Concentration (Cmax) of Durvalumab
Description: Serum samples were collected from the participants at the defined timepoints. Cmax was determined using standard non-compartmental methods.
Time Frame: Pre-infusion and post-infusion on Cycle 1 Day 1, Cycle 1 Day 8, Cycle 1 Day 15, pre-infusion and post-infusion on Cycle 2 Day 1, pre-infusion and post-infusion in Cycle 3, 4, 6, 8, 10 and 12
Population: The pharmacokinetic (PK) analysis set included all participants who received at least 1 dose of study treatment per the clinical study protocol (CSP) for whom any post-dose data were available who did not violate or deviate from the CSP in ways that would significantly affect the PK analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/ milliliter (mcg/mL)
Arm/Group | Arm A (>= 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm A (>= 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 7 | 11 | 3 | 8
micrograms/ milliliter (mcg/mL) | 363 (58.0) | 865 (36.0) | 275 (135) | 612 (34.2)

2. Primary Outcome: Dose-Finding Phase: Minimum Serum Concentration (Cmin) of Durvalumab
Description: Serum samples were collected from the participants at the defined timepoints. Cmin was determined using standard non-compartmental methods.
Time Frame: as for outcome 1
Population: The PK analysis set included all participants who received at least 1 dose of study treatment per the CSP for whom any post-dose data were available who did not violate or deviate from the CSP in ways that would significantly affect the PK analysis. Only data from the participants analyzed were reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Arm A (>= 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm A (>= 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 6 | 8 | 3 | 4
mcg/mL | 48.6 (104) | 169 (28.5) | 21.7 (34.6) | 118 (45.4)

3. Primary Outcome: Dose-Finding Phase: Area Under the Serum Concentration-Time Curve (AUC) From Zero to 14 (AUC 0-14) of Durvalumab
Description: Serum samples were collected from the participants at the defined timepoints. AUC (0-14) was determined using standard non-compartmental methods.
Time Frame: Pre-infusion and post-infusion on Cycle 1 Day 1 and Cycle 1 Day 8
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*mcg/mL
Arm/Group | Arm A (>= 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm A (>= 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 7 | 9 | 3 | 6
day*mcg/mL | 2650 (61.5) | 5660 (17.7) | 1830 (54.7) | 3720 (46.9)

4. Primary Outcome: Dose-Finding Phase: AUC From Zero to 28 (AUC 0-28) of Durvalumab
Description: Serum samples were collected from the participants at the defined timepoints. AUC (0-28) was determined using standard non-compartmental methods.
Time Frame: Pre-infusion and post-infusion on Cycle 1 Day 1, Cycle 1 Day 8, and Cycle 1 Day 15
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*mcg/mL
Arm/Group | Arm A (>= 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm A (>= 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 6 | 8 | 3 | 4
day*mcg/mL | 3290 (50.1) | 8790 (13.5) | 2500 (55.4) | 6380 (40.1)

5. Primary Outcome: Dose-Finding Phase: Time to Cmax (Tmax) of Durvalumab
Description: Serum samples were collected from the participants at the defined timepoints. Tmax was determined using standard non-compartmental methods.
Time Frame: as for outcome 1
Population: The PK analysis set included all participants who received at least 1 dose of study treatment per the CSP for whom any post-dose data were available who did not violate or deviate from the CSP in ways that would significantly affect the PK analysis.
Measure: Median (Full Range); unit: days
Arm/Group | Arm A (>= 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm A (>= 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 7 | 11 | 3 | 8
days | 0.094 [0.09 to 0.10] | 0.087 [0.00 to 0.14] | 0.09 [0.09 to 6.94] | 0.087 [0.08 to 0.09]

6. Primary Outcome: Dose-Finding Phase: Apparent Terminal Elimination Half-life Associated With the Terminal Slope of the Semi-logarithmic Concentration Time Curve (t½λz) of Durvalumab
Description: Serum samples were collected from the participants at the defined timepoints. T½λz was determined using standard non-compartmental methods.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | Arm A (>= 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm A (>= 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 6 | 6 | 1 | 2
days | 16.7 (47.1) | 25.3 (56.5) | 8.26 (NA) — NA indicates geometric coefficient of variation was not calculated for 1 participant. | 15.6 (23.3)

7. Primary Outcome: Dose-Finding Phase: Dose-Normalized AUC (0-14) (AUC [0-14]/D) of Durvalumab
Description: Serum samples were collected from the participants at the defined timepoints. AUC(0-14)/D was determined using standard non-compartmental methods.
Time Frame: Pre-infusion and post-infusion on Cycle 1 Day 1 and Cycle 1 Day 8
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (day*mcg/mL)/(mg/kg)
Arm/Group | Arm A (>= 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm A (>= 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 7 | 9 | 3 | 6
(day*mcg/mL)/(mg/kg) | 132 (61.5) | 189 (17.7) | 91.6 (54.7) | 124 (46.9)

8. Primary Outcome: Dose-Finding Phase: Dose-Normalized AUC (0-28) (AUC [0-28]/D) of Durvalumab
Description: Serum samples were collected from the participants at the defined timepoints. AUC(0-28)/D was determined using standard non-compartmental methods.
Time Frame: Pre-infusion and post-infusion on Cycle 1 Day 1, Cycle 1 Day 8, and Cycle 1 Day 15
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (day*mcg/mL)/(mg/kg)
Arm/Group | Arm A (>= 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm A (>= 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 6 | 8 | 3 | 4
(day*mcg/mL)/(mg/kg) | 164 (50.1) | 293 (13.5) | 125 (55.4) | 213 (40.1)

9. Primary Outcome: Dose-Finding Phase: Dose-Normalized Cmax (Cmax/D) of Durvalumab
Description: Serum samples were collected from the participants at the defined timepoints. Cmax/D was determined using standard non-compartmental methods.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (mcg/mL)/(mg/kg)
Arm/Group | Arm A (>= 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm A (>= 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 7 | 11 | 3 | 8
(mcg/mL)/(mg/kg) | 18.1 (58.0) | 28.8 (36.0) | 13.7 (135) | 20.4 (34.2)

10. Primary Outcome: Dose-Finding Phase: Cmax of Tremelimumab
Description: as for outcome 1
Time Frame: Pre-infusion and post-infusion on Cycle 2 Day 1, Cycle 2 Day 8, Cycle 2 Day 15, pre-infusion and post-infusion in Cycle 3, 4, and 5
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Arm A (>= 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm A (>= 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 6 | 8 | 3 | 4
mcg/mL | 19.1 (73.3) | 24.5 (44.7) | 39.2 (68.8) | 23.0 (31.7)

11. Primary Outcome: Dose-Finding Phase: Cmin of Tremelimumab
Description: as for outcome 2
Time Frame: as for outcome 10
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Arm A (>= 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm A (>= 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 2 | 4 | 0 | 3
mcg/mL | 3.71 (3.75) | 3.45 (29.2) |  | 3.03 (50.3)

12. Primary Outcome: Dose-Finding Phase: (AUC 0-14) of Tremelimumab
Description: as for outcome 3
Time Frame: Pre-infusion and post-infusion on Cycle 2 Day 1, and Cycle 2 Day 8
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*mcg/mL
Arm/Group | Arm A (>= 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm A (>= 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 5 | 7 | 2 | 4
day*mcg/mL | 127 (47.3) | 160 (35.6) | 165 (7.00) | 149 (20.1)

13. Primary Outcome: Dose-Finding Phase: (AUC 0-28) of Tremelimumab
Description: as for outcome 4
Time Frame: Pre-infusion and post-infusion on Cycle 2 Day 1, Cycle 2 Day 8, and Cycle 2 Day 15
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*mcg/mL
Arm/Group | Arm A (>= 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm A (>= 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 2 | 4 | 0 | 3
day*mcg/mL | 235 (11.2) | 205 (22.9) |  | 208 (14.8)

14. Primary Outcome: Dose-Finding Phase: Tmax of Tremelimumab
Description: as for outcome 5
Time Frame: as for outcome 10
Population: as for outcome 2
Measure: Median (Full Range); unit: days
Arm/Group | Arm A (>= 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm A (>= 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 6 | 8 | 3 | 4
days | 0.046 [0.04 to 0.08] | 0.051 [0.04 to 0.07] | 0.040 [0.04 to 0.05] | 0.046 [0.04 to 0.18]

15. Primary Outcome: Dose-Finding Phase: T½λz of Tremelimumab
Description: as for outcome 6
Time Frame: as for outcome 10
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | Arm A (>= 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm A (>= 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 2 | 3 | 0 | 2
days | 16.8 (5.27) | 18.7 (20.5) |  | 31.6 (86.0)

16. Primary Outcome: Dose-Finding Phase: AUC (0-14)/D of Tremelimumab
Description: as for outcome 7
Time Frame: Pre-infusion and post-infusion on Cycle 2 Day 1 and Cycle 2 Day 8
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (day*mcg/mL)/(mg/kg)
Arm/Group | Arm A (>= 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm A (>= 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 5 | 7 | 2 | 4
(day*mcg/mL)/(mg/kg) | 127 (47.3) | 160 (35.6) | 165 (7.00) | 149 (20.1)

17. Primary Outcome: Dose-Finding Phase: AUC (0-28)/D of Tremelimumab
Description: as for outcome 8
Time Frame: Pre-infusion and post-infusion on Cycle 2 Day 1, Cycle 2 Day 8, and Cycle 2 Day 15
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (day*mcg/mL)/(mg/kg)
Arm/Group | Arm A (>= 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm A (>= 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 2 | 4 | 0 | 3
(day*mcg/mL)/(mg/kg) | 235 (11.2) | 205 (22.9) |  | 208 (14.8)

18. Primary Outcome: Dose-Finding Phase: Cmax/D of Tremelimumab
Description: as for outcome 9
Time Frame: as for outcome 10
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (mcg/mL)/(mg/kg)
Arm/Group | Arm A (>= 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm A (>= 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 6 | 8 | 3 | 4
(mcg/mL)/(mg/kg) | 19.1 (73.3) | 24.5 (44.7) | 39.2 (68.8) | 23.0 (31.7)

19. Primary Outcome: Dose-Finding Phase: Number of Participants With Adverse Events (AE), Serious AE (SAE), AE Leading to Discontinuation of Durvalumab and Tremelimumab, AE of Special Interest (AESI) or AE of Possible Interest (AEPI) Related to Durvalumab and Tremelimumab
Description: An AE was defined as any untoward medical occurrence in a participant temporally associated with the use of study treatment, whether or not considered related to the study treatment. SAEs were any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. Some AEs and higher-level terms were considered AESI or AEPIs and this list of categories were provided by the patient safety team.
Time Frame: From Day 1 up to 15 months
Population: The Safety analysis set included all participants who received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (>= 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm A (>= 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 7 | 11 | 3 | 8
Participants
  Any AE | 6 | 11 | 3 | 7
  Any SAE | 1 | 1 | 0 | 1
  AE leading to discontinuation of Durvalumab | 0 | 0 | 0 | 0
  AE leading to discontinuation of Tremelimumab | 0 | 1 | 0 | 0
  AESIs or AEPIs related to Durvalumab | 1 | 4 | 0 | 2
  AESIs or AEPIs related to Tremelimumab | 0 | 2 | 0 | 1

20. Primary Outcome: Dose-Expansion Phase Only: Objective Response Rate (ORR)
Description: ORR as per RECIST 1.1 was defined as the percentage of participants with at least 1 investigator-assessed visit response of complete response (CR) or partial response (PR) that was subsequently confirmed on another scan not less than 4 weeks after visit observed response. CR was defined as disappearance of all target lesions (TLs), any pathological lymph nodes selected as TLs with reduction in short axis to < 10 millimeter (mm). PR was defined as at least a 30% decrease in the sum of diameters of TLs, with reference to baseline sum of diameters as long as criteria for PD are not met.
Time Frame: From first dose of study treatment until death or up to approximately 4 years (clinical DCO of 20 Apr 2023)
Population: The evaluable for response analysis set is the subset of participants in the FAS who had measurable disease (as per RECIST 1.1) at baseline and had at least 1 follow-up scan measuring all required target lesions and had been followed for at least 3 cycles or measurable disease (as per RECIST 1.1) at baseline and progressed or died in the absence of a follow-up scan.
Measure: Number; unit: percentage of participants
Arm/Group | SARCOMA: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | STO: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 11 | 9
percentage of participants | 0 | 11.1

21. Primary Outcome: Dose-Expansion Phase Only: Duration of Response (DOR)
Description: Duration of response was the time from the first documentation of CR/PR (which was subsequently confirmed) until the date of documented progression, or death which coincides with the progression free survival (PFS) endpoint. For participants who did not progress following a response, the DOR was censored during the PFS censoring time. It was calculated using Kaplan-Meier technique.
Time Frame: From first dose of study treatment until death or up to approximately 4 years (clinical DCO of 20 Apr 2023)
Population: The evaluable for response analysis set is the subset of participants in the FAS who had measurable disease (as per RECIST 1.1) at baseline and had at least 1 follow-up scan measuring all required target lesions and had been followed for at least 3 cycles or measurable disease (as per RECIST 1.1) at baseline and progressed or died in the absence of a follow-up scan. Only responders were included in this analysis.
Measure: Median (Full Range); unit: months
Arm/Group | SARCOMA: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | STO: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 0 | 1
months |  | 10.8 [10.8 to 10.8]

22. Primary Outcome: Dose-Expansion Phase Only: Best Objective Response (BOR)
Description: BOR was calculated based on the overall visit responses from each RECIST 1.1 assessment. Categorization of BOR for solid tumors were based on RECIST 1.1 using the following response categories: CR, PR, stable disease (SD), progression of disease (PD), and not evaluable (NE). CR: disappearance of all TLs. Any pathological lymph nodes selected as TLs had a reduction in short axis to <10 mm. PR: 30% decrease in the sum of diameters of TLs. SD: Neither sufficient decrease in sum of diameters to qualify for PR nor sufficient increased to qualify for PD. PD: >= 20 % increase in the sum of diameters to TLs and an increase of >= 5 mm. NE: Only relevant if any of the TLs were not assessed or NE or had a lesion intervention at visit. Non-CR/Non-PD: Persistence of 1+ non-target lesion (s). Non-CR/non-PD was relevant to participants who did not have measurable disease at baseline.
Time Frame: From first dose of study treatment until death or up to approximately 4 years (clinical DCO of 20 Apr 2023)
Population: The FAS included all participants who were assigned to treatment and received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | SARCOMA: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | STO: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 11 | 10
Participants
  CR | 0 | 0
  PR | 0 | 1
  Unconfirmed complete or partial response | 0 | 0
  SD >= 7 weeks | 1 | 1
  PD | 9 | 7
  Not evaluable | 1 | 1

23. Primary Outcome: Dose-Expansion Phase Only: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants who achieved a BOR of unconfirmed CR or PR, respectively, or who had SD. CR was defined as disappearance of all TLs, any pathological lymph nodes selected as TLs with reduction in short axis to < 10 mm. PR was defined as at least a 30% decrease in the sum of diameters of TLs, with reference to baseline sum of diameters as long as criteria for PD are not met. SD: Neither sufficient decrease in sum of diameters to qualify for PR nor sufficient increased to qualify for PD.
Time Frame: At 16 and 24 Weeks
Population: The FAS included all participants who were assigned to treatment and received at least 1 dose of study treatment. Only participants who achieved a BOR were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | SARCOMA: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | STO: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 11 | 10
percentage of participants
  Week 16 | 9.1 | 10.0
  Week 24 | 9.1 | 10.0

24. Primary Outcome: Dose-Expansion Phase Only: PFS
Description: PFS as per RECIST 1.1 was defined as the time from the date of first dose of study treatment until the date of objective disease progression or death by any cause in the absence of progression, regardless of whether the participant withdrew from study therapy or received another anti-cancer therapy prior to progression (date of PFS event or censoring - date of first dose + 1). Confidence interval was calculated using Kaplan-Meier technique.
Time Frame: From first dose of study treatment until death or up to approximately 4 years (clinical DCO of 20 Apr 2023)
Population: The FAS included all participants who were assigned to treatment and received at least 1 dose of study treatment.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | SARCOMA: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | STO: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 11 | 10
months | 1.7 [1.58 to 1.91] | 1.7 [0.89 to 2.76]

25. Primary Outcome: Dose-Expansion Phase Only: Overall Survival (OS)
Description: OS was defined as the time from the date of first dose of study treatment until death due to any cause regardless of whether the patient withdraws from study treatment or received another anti-cancer therapy (i.e date of death or censoring - date of first dose + 1).
Time Frame: From first dose of study treatment until death or up to approximately 4 years (clinical DCO of 20 Apr 2023)
Population: The FAS included all participants who were assigned to treatment and received at least 1 dose of study treatment.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | SARCOMA: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | STO: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 11 | 10
months | 6.6 [2.2 to 15.8] | 6.9 [3.2 to NA] — NA indicates higher inter-quartile range not reached.

26. Primary Outcome: Dose-Expansion Phase Only: Survival Rate at 12 Months and 24 Months
Description: Survival rates were defined as the Kaplan-Meier estimate of OS at 12 and 24 months.
Time Frame: At 12 and 24 Weeks
Population: The FAS included all participants who were assigned to treatment and received at least 1 dose of study treatment.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | SARCOMA: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | STO: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 11 | 10
percentage of participants
  12 Months | 25.6 [6.27 to 51.10] | 40.0 [15.94 to 63.31]
  24 Months | NA [NA to NA] — NA indicated survival rate not reached for 24 months at this DCO. | 30.0 [9.74 to 53.67]

27. Secondary Outcome: Dose-Expansion Phase: Cmax of Durvalumab
Description: as for outcome 1
Time Frame: Pre-infusion and post-infusion on Cycle 1 Day 1, Cycle 1 Day 8, Cycle 1 Day 15, pre-infusion and post-infusion on Cycle 2 Day 1, pre-infusion and post-infusion in Cycle 3, 4, 8, and 12
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | SARCOMA: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | STO: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 11 | 10
mcg/mL | 606 (27.7) | 595 (14.2)

28. Secondary Outcome: Dose-Expansion Phase: Cmin of Durvalumab
Description: as for outcome 2
Time Frame: as for outcome 27
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | SARCOMA: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | STO: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 9 | 5
mcg/mL | 108 (29.6) | 78.3 (94.1)

29. Secondary Outcome: Dose-Expansion Phase: AUC (0-14) of Durvalumab
Description: as for outcome 3
Time Frame: Pre-infusion and post-infusion on Cycle 1 Day 1 and Cycle 1 Day 8
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*mcg/mL
Arm/Group | SARCOMA: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | STO: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 10 | 9
day*mcg/mL | 4240 (23.2) | 3900 (20.0)

30. Secondary Outcome: Dose-Expansion Phase: AUC (0-28) of Durvalumab
Description: as for outcome 4
Time Frame: Pre-infusion and post-infusion on Cycle 1 Day 1, Cycle 1 Day 8, and Cycle 1 Day 15
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*mcg/mL
Arm/Group | SARCOMA: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | STO: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 9 | 5
day*mcg/mL | 6400 (23.7) | 5880 (25.2)

31. Secondary Outcome: Dose-Expansion Phase: Tmax of Durvalumab
Description: as for outcome 5
Time Frame: as for outcome 27
Population: as for outcome 5
Measure: Median (Full Range); unit: days
Arm/Group | SARCOMA: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | STO: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 11 | 10
days | 0.049 [0.04 to 0.09] | 0.051 [0.04 to 0.08]

32. Secondary Outcome: Dose-Expansion Phase: T½λz of Durvalumab
Description: as for outcome 6
Time Frame: as for outcome 27
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | SARCOMA: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | STO: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 8 | 5
days | 17.4 (26.2) | 14.2 (48.6)

33. Secondary Outcome: Dose-Expansion Phase: AUC (0-14)/D of Durvalumab
Description: Serum samples were collected from the participants at the defined timepoints. AUC (0-14)/D was determined using standard non-compartmental methods.
Time Frame: Pre-infusion and post-infusion on Cycle 1 Day 1 and Cycle 1 Day 8
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (day*mcg/mL)/(mg/kg)
Arm/Group | SARCOMA: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | STO: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 10 | 9
(day*mcg/mL)/(mg/kg) | 141 (23.2) | 130 (20.0)

34. Secondary Outcome: Dose-Expansion Phase: AUC (0-28)/D of Durvalumab
Description: Serum samples were collected from the participants at the defined timepoints. AUC (0-28)/D was determined using standard non-compartmental methods.
Time Frame: Pre-infusion and post-infusion on Cycle 1 Day 1, Cycle 1 Day 8, and Cycle 1 Day 15
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (day*mcg/mL)/(mg/kg)
Arm/Group | SARCOMA: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | STO: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 9 | 5
(day*mcg/mL)/(mg/kg) | 213 (23.7) | 196 (25.2)

35. Secondary Outcome: Dose-Expansion Phase: Cmax/D of Durvalumab
Description: as for outcome 9
Time Frame: as for outcome 27
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (mcg/mL)/(mg/kg)
Arm/Group | SARCOMA: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | STO: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 11 | 10
(mcg/mL)/(mg/kg) | 20.2 (27.7) | 19.8 (14.2)

36. Secondary Outcome: Dose-Expansion Phase: Cmax of Tremelimumab
Description: as for outcome 1
Time Frame: Pre-infusion and post-infusion on Cycle 1 Day 1, Cycle 1 Day 8, Cycle 1 Day 15, pre-infusion and post-infusion on Cycle 2 Day 1, Cycle 3 Day 1 pre-infusion and post-infusion on Cycle 4
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | SARCOMA: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | STO: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 10 | 10
mcg/mL | 29.2 (86.0) | 23.2 (18.8)

37. Secondary Outcome: Dose-Expansion Phase: Cmin of Tremelimumab
Description: as for outcome 2
Time Frame: as for outcome 36
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | SARCOMA: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | STO: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 9 | 6
mcg/mL | 3.91 (41.7) | 3.40 (66.2)

38. Secondary Outcome: Dose-Expansion Phase: AUC (0-14) of Tremelimumab
Description: as for outcome 3
Time Frame: Pre-infusion and post-infusion on Cycle 1 Day 1 and Cycle 1 Day 8
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*mcg/mL
Arm/Group | SARCOMA: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | STO: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 10 | 8
day*mcg/mL | 183 (65.9) | 150 (11.8)

39. Secondary Outcome: Dose-Expansion Phase: AUC (0-28) of Tremelimumab
Description: as for outcome 4
Time Frame: Pre-infusion and post-infusion on Cycle 1 Day 1, Cycle 1 Day 8, and Cycle 1 Day 15
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*mcg/mL
Arm/Group | SARCOMA: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | STO: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 9 | 6
day*mcg/mL | 270 (58.1) | 228 (12.4)

40. Secondary Outcome: Dose-Expansion Phase: Tmax of Tremelimumab
Description: as for outcome 5
Time Frame: as for outcome 36
Population: as for outcome 2
Measure: Median (Full Range); unit: days
Arm/Group | SARCOMA: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | STO: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 10 | 10
days | 0.049 [0.04 to 0.06] | 0.052 [0.04 to 0.07]

41. Secondary Outcome: Dose-Expansion Phase: T½λz of Tremelimumab
Description: as for outcome 6
Time Frame: as for outcome 36
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | SARCOMA: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | STO: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 7 | 6
days | 15.9 (26.2) | 15.6 (40.4)

42. Secondary Outcome: Dose-Expansion Phase: AUC (0-14)/D of Tremelimumab
Description: as for outcome 33
Time Frame: Pre-infusion and post-infusion on Cycle 1 Day 1 and Cycle 1 Day 8
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (day*mcg/mL)/(mg/kg)
Arm/Group | SARCOMA: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | STO: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 10 | 8
(day*mcg/mL)/(mg/kg) | 183 (65.9) | 150 (11.8)

43. Secondary Outcome: Dose-Expansion Phase: AUC (0-28)/D of Tremelimumab
Description: as for outcome 34
Time Frame: Pre-infusion and post-infusion on Cycle 1 Day 1, Cycle 1 Day 8, and Cycle 1 Day 15
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (day*mcg/mL)/(mg/kg)
Arm/Group | SARCOMA: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | STO: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 9 | 6
(day*mcg/mL)/(mg/kg) | 270 (58.1) | 228 (12.4)

44. Secondary Outcome: Dose-Expansion Phase: Cmax/D of Tremelimumab
Description: as for outcome 9
Time Frame: as for outcome 36
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (mcg/mL)/(mg/kg)
Arm/Group | SARCOMA: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | STO: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 10 | 10
(mcg/mL)/(mg/kg) | 29.2 (86.0) | 23.2 (18.8)

45. Secondary Outcome: Dose-Finding Phase: Percentage of Participants Who Developed Detectable Anti-Drug Antibodies (ADAs)
Description: ADA prevalence was defined as the percentage of participants with positive ADA result at any time, baseline or post-baseline. Persistently positive was defined as having at least 2 post-baseline ADA positive measurements with at least 16 weeks (112 days) between the first and last positive measurements, or an ADA positive result at the last available assessment. Transiently positive was defined as having at least 1 post-baseline ADA positive measurement and not fulfilling the conditions for persistently positive.
Time Frame: Pre-infusion on Cycle 1 Day 1 and Cycle 3 Day 1 (durvalumab and tremelimumab), pre-infusion on Cycle 2 Day 1, Cycle 5 Day 1 and Cycle 8 Day 1 for tremelimumab
Population: The ADA analysis set included all participants who received at least 1 dose of study treatment per the CSP for whom baseline, and any post-dose data were available were included in the ADA analysis set. Only data from the participants analyzed were reported.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A (>= 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm A (>= 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 4 | 3 | 1 | 1
percentage of participants
  Durvalumab, ADA positive at any visit | 25 | 0 | 0 | 0
  Durvalumab, Persistently positive | 0 | 0 | 0 | 0
  Durvalumab, Transiently positive | 0 | 0 | 0 | 0
  Tremelimumab, ADA positive at any visit | 0 | 0 | 0 | 0
  Tremelimumab, Persistently positive | 0 | 0 | 0 | 0
  Tremelimumab, Transiently positive | 0 | 0 | 0 | 0

46. Secondary Outcome: Dose-Expansion Phase: Percentage of Participants Who Developed Detectable ADAs
Description: ADA prevalence was defined as the percentage of participants with positive ADA result at any time, baseline or post-baseline. Persistently positive was defined as having at least 2 post-baseline ADA positive measurements with at least 16 weeks (112 days) between the first and last positive measurements, or an ADA positive result at the last available assessment. The category includes participants meeting these criteria who are ADA positive at baseline. Transiently positive was defined as having at least 1 post-baseline ADA positive measurement and not fulfilling the conditions for persistently positive. The category includes participants meeting these criteria who are ADA positive at baseline.
Time Frame: Pre-infusion on Cycle 1 Day 1 and Cycle 3 Day 1 (durvalumab and tremelimumab) and random sample on Cycle 7 Day 1 for tremelimumab
Population: The ADA analysis set included all participants who received at least 1 dose of study treatment per the CSP for whom baseline, and any post-dose data were available were included in the ADA analysis set.
Measure: Number; unit: percentage of participants
Arm/Group | SARCOMA: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | STO: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 4 | 5
percentage of participants
  Durvalumab, ADA positive at any visit | 0 | 20
  Durvalumab, Persistently positive | 0 | 0
  Durvalumab, Transiently positive | 0 | 0
  Tremelimumab, ADA positive at any visit | 0 | 0
  Tremelimumab, Persistently positive | 0 | 0
  Tremelimumab, Transiently positive | 0 | 0

47. Secondary Outcome: Number of Participants With Individual Antibody Titer Measurement
Description: Blood samples were planned to be collected for vaccine antibody titer measurements before and after planned routine immunization.
Time Frame: Pre-infusion on Cycle 1 Day 1 and Cycle 4 Day 1 for durvalumab, pre-infusion on Cycle 1 Day 1, pre-infusion on Cycle 3, 4, and 8 Day 1 for tremelimumab (dose-expansion)
Population: Participants who has a baseline titer collected and who has subsequent samples following a routine childhood immunization were included. As no participants received a routine immunization during the study, no additional samples were collected, hence no data analysed.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (>= 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm A (>= 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | SARCOMA: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | STO: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 7 | 11 | 3 | 8 | 11 | 10
Participants | 0 | 0 | 0 | 0 | 0 | 0

48. Secondary Outcome: Median Percent Change From Baseline of Cluster of Differentiation 4+ (CD4+), CD8+, B Cells, Natural Killer (NK) Cells, and T-cell Activation With Ki67
Description: Blood samples were collected at indicated timepoints for flow cytometry assessment. Cycle (C) and Day (D). Data collected for the flow cytometry analysis from the participants enrolled in both the dose finding and dose expansion phase were analyzed in the context of the dosing regimen received, to determine any potential differences in the immune response based on the durvalumab dose.
Time Frame: Pre-dose Cycle 1 Day 8, pre-dose Cycle 2 Day 1, Cycle 2 Day 8, pre-dose Cycle 3 Day 1 (Dose-finding); Pre-dose Cycle 1 Day 1, Cycle 1 Day 8, pre-dose Cycle 2 Day 1 (Dose-expansion)
Population: Participants who received the Durvalumab + tremelimumab combination who had a pre-treatment sample collected on Day 1 and a repeat sample on Day 8 were included. As the weight of the participant was not believed to impact the immune response, it was determined that aggregating the data by dosing regimen rather than by weight group, was considered acceptable for this particular analysis.
Measure: Median (Inter-Quartile Range); unit: percentage of cells per cubic millimeter
Groups:
- Dose Expansion: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg: Participants from cohort SARCOMA and STO, who were administered durvalumab 30 mg/kg IV in combination with tremelimumab 1 mg/kg IV in Cycles 1-4 every 28 days. From Cycle 5, onwards participants were administered durvalumab 30 mg/kg every 28 days until clinical or confirmed disease progression or until any of other discontinuation criterion was met, whichever occurred first.
- Dose Finding: Durvalumab 20 mg/kg + Tremelimumab 1mg/kg: Participants who weighed >= 35 kg in Arm A and < 35 kg in Arm B were administered durvalumab 20 mg/kg IV in Cycle 1 followed by durvalumab in combination with tremelimumab 1 mg/kg IV in Cycles 2-5 every 28 days. From Cycle 6, onwards participants were administered durvalumab 20 mg/kg every 28 days until clinical or confirmed disease progression or until any of other discontinuation criterion was met, whichever occurred first.
- Dose Finding: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg: Participants who weighed >= 35 kg in Arm A and < 35 kg in Arm B were administered durvalumab 30 mg/kg IV in Cycle 1 followed by durvalumab in combination with tremelimumab 1 mg/kg IV for Cycles 2-5 every 28 days. From Cycle 6, onwards participants were administered durvalumab 20 mg/kg every 28 days until clinical or confirmed disease progression or until any of other discontinuation criterion was met, whichever occurred first.
Arm/Group | Dose Expansion: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | Dose Finding: Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Dose Finding: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
Number analyzed (Participants) | 12 | 7 | 7
percentage of cells per cubic millimeter
  T cells CD4+ Ki67; C1D8: number analyzed (Participants) | 12 | 0 | 0
  T cells CD4+ Ki67; C1D8 | 112.8 [69.2 to 352.5] |  |
  T cells CD4+ Ki67; C2D1: number analyzed (Participants) | 8 | 7 | 6
  T cells CD4+ Ki67; C2D1 | 10.3 [-45.8 to 57.6] | 16.7 [-24.0 to 66.7] | -25.8 [-43.8 to 37.8]
  T cells CD4+ Ki67; C2D8: number analyzed (Participants) | 0 | 6 | 5
  T cells CD4+ Ki67; C2D8 |  | 153.1 [58.0 to 925.0] | 118.2 [65.1 to 215.0]
  T cells CD4+ Ki67; C3D1: number analyzed (Participants) | 0 | 2 | 3
  T cells CD4+ Ki67; C3D1 |  | -33.4 [-48.0 to -18.8] | 21.9 [-31.4 to 81.3]
  T cells CD8+ Ki67; C1D8: number analyzed (Participants) | 7 | 0 | 0
  T cells CD8+ Ki67; C1D8 | 20.0 [-25.0 to 88.9] |  |
  T cells CD8+ Ki67; C2D1: number analyzed (Participants) | 5 | 6 | 6
  T cells CD8+ Ki67; C2D1 | -20.0 [-70.8 to 117.5] | 133.3 [-9.9 to 431.3] | -62.1 [-67.5 to 173.3]
  T cells CD8+ Ki67; C2D8: number analyzed (Participants) | 0 | 5 | 5
  T cells CD8+ Ki67; C2D8 |  | 66.7 [-35.2 to 900.0] | -40.0 [-57.0 to 318.3]
  T cells CD8+ Ki67; C3D1: number analyzed (Participants) | 0 | 1 | 3
  T cells CD8+ Ki67; C3D1 |  | 0.0 [0.0 to 0.0] | -55.4 [-73.0 to 200.0]
  T cells CD4+; C1D8: number analyzed (Participants) | 12 | 0 | 0
  T cells CD4+; C1D8 | -12.5 [-20.5 to 2.9] |  |
  T cells CD4+; C2D1: number analyzed (Participants) | 9 | 7 | 7
  T cells CD4+; C2D1 | 10.1 [-15.2 to 26.2] | 6.1 [-20.2 to 45.7] | 9.2 [-16.6 to 34.9]
  T cells CD4+; C2D8: number analyzed (Participants) | 0 | 6 | 6
  T cells CD4+; C2D8 |  | 12.8 [-6.5 to 63.8] | 16.1 [-13.2 to 52.7]
  T cells CD4+; C3D1: number analyzed (Participants) | 0 | 2 | 4
  T cells CD4+; C3D1 |  | -12.3 [-32.6 to 8.0] | 23.0 [6.3 to 39.9]
  T cells CD8+; C1D8: number analyzed (Participants) | 12 | 0 | 0
  T cells CD8+; C1D8 | -23.3 [-37.8 to -10.3] |  |
  T cells CD8+; C2D1: number analyzed (Participants) | 9 | 7 | 7
  T cells CD8+; C2D1 | 3.6 [-30.2 to 23.1] | 40.4 [-18.2 to 59.2] | 10.6 [-15.6 to 50.6]
  T cells CD8+; C2D8: number analyzed (Participants) | 0 | 6 | 6
  T cells CD8+; C2D8 |  | 30.1 [-14.6 to 60.9] | 13.8 [-18.0 to 71.2]
  T cells CD8+; C3D1: number analyzed (Participants) | 0 | 2 | 4
  T cells CD8+; C3D1 |  | -8.3 [-24.5 to 7.9] | 0.6 [-5.5 to 2.6]
  B cells; C1D8: number analyzed (Participants) | 12 | 0 | 0
  B cells; C1D8 | -29.2 [-40.6 to -24.7] |  |
  B cells; C2D1: number analyzed (Participants) | 9 | 7 | 7
  B cells; C2D1 | 6.2 [-3.1 to 56.9] | 27.2 [-1.5 to 650.0] | -12.0 [-22.0 to 128.0]
  B cells; C2D8: number analyzed (Participants) | 0 | 6 | 6
  B cells; C2D8 |  | 20.6 [-4.8 to 1543.8] | -8.2 [-26.2 to 43.1]
  B cells; C3D1: number analyzed (Participants) | 0 | 2 | 4
  B cells; C3D1 |  | -2.5 [-8.6 to 3.6] | 15.7 [-24.4 to 42.1]
  NK cells; C1D8: number analyzed (Participants) | 12 | 0 | 0
  NK cells; C1D8 | -30.1 [-39.7 to 15.2] |  |
  NK cells; C2D1: number analyzed (Participants) | 9 | 7 | 7
  NK cells; C2D1 | -25.8 [-49.2 to 55.3] | 31.0 [-1.1 to 59.6] | 32.2 [14.3 to 56.8]
  NK cells; C2D8: number analyzed (Participants) | 0 | 6 | 6
  NK cells; C2D8 |  | 7.4 [-28.1 to 75.9] | 47.4 [22.2 to 55.6]
  NK cells; C3D1: number analyzed (Participants) | 0 | 2 | 4
  NK cells; C3D1 |  | 25.9 [-9.6 to 61.4] | 43.7 [-26.9 to 77.2]

ADVERSE EVENTS:
Time Frame: From first dose of study treatment up to approximately 4 years (clinical DCO of 20 Apr 2023)
Description: The safety analysis set included all participants who received any amount of study treatment.
Arm/Group | Arm A (>= 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm A (>= 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg | Arm B (< 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | SARCOMA: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg | STO: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg
All-Cause Mortality (participants affected / at risk) | 6/7 | 8/11 | 3/3 | 7/8 | 8/11 | 7/10
Serious Adverse Events (participants affected / at risk) | 1/7 | 1/11 | 0/3 | 1/8 | 6/11 | 3/10
Other Adverse Events (participants affected / at risk) | 6/7 | 11/11 | 3/3 | 7/8 | 8/11 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (>= 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg (N=7) | Arm A (>= 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg (N=11) | Arm B (< 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg (N=3) | Arm B (< 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg (N=8) | SARCOMA: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg (N=11) | STO: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg (N=10)
Transverse sinus thrombosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (>= 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg (N=7) | Arm A (>= 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg (N=11) | Arm B (< 35 kg): Durvalumab 20 mg/kg + Tremelimumab 1mg/kg (N=3) | Arm B (< 35 kg): Durvalumab 30 mg/kg + Tremelimumab 1mg/kg (N=8) | SARCOMA: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg (N=11) | STO: Durvalumab 30 mg/kg + Tremelimumab 1mg/kg (N=10)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Amputation stump pain (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anosmia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 4 (5) | 0 (0) | 2 (7) | 1 (1) | 2 (3)
Horner's syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Glycosuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocyturia (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 3 (4) | 1 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin depigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (5) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (3) | 1 (1) | 1 (1) | 4 (5) | 3 (4)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 7 (10) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (5) | 2 (3) | 0 (0) | 3 (6) | 2 (2) | 2 (6)
Asthenia (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Papillitis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 1 (2) | 0 (0) | 2 (2) | 6 (9) | 4 (5)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bed bug infestation (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (6) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 4 (5) | 1 (1) | 1 (1) | 2 (4) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (4) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bicarbonate decreased (Investigations) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram T wave abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (5) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embryonal rhabdomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/99/NCT03837899/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-19): https://cdn.clinicaltrials.gov/large-docs/99/NCT03837899/SAP_001.pdf